CLINICAL TRIAL: NCT00605098
Title: Pharmacokinetics of the Tablet Formulation of Lopinavir/r as Standard and Increased Dosage During Pregnancy in HIV-infected Women
Brief Title: Pharmacokinetics of the Tablet Formulation of Lopinavir/r as Standard and Increased Dosage During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Marilia Santini de Oliveira, Medical doctor, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PK-LPV 01
Record Dates: First submitted 2008-01-07; First posted 2008-01-30 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: HIV; Pregnancy; Vertical disease transmission; Pharmacokinetics; HIV seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Lopinavir / ritonavir
- 2 (Experimental)
  Interventions: Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Lopinavir / ritonavir — Lopinavir/r (200/50 mg, 2 tablets every 12 hours) plus two nucleoside analogs, starting at any time between 14 and 30 weeks of gestation and maintained for at least 6 weeks after delivery.
  Other Names: Kaletra
  Arms: 1
Drug: Lopinavir/ritonavir — Lopinavir/r (200/50 mg, 2 tablets every 12 hours) plus two nucleoside analogs, starting at any time between 14 and 30 weeks of gestation, increase the lopinavir/r dosage (200/50 mg, 3 tablets every 12 hours) in the third trimester (from 25 weeks on), and return to standard dose(200/50 mg, 2 tablets every 12 hours)for at least 6 weeks after delivery.
  Other Names: Kaletra
  Arms: 2

SUMMARY:
This is a multicenter, open, prospective and randomized study aimed at evaluating the pharmacokinetics of the tablet formulation of lopinavir/r administered in combination with two nucleoside analogs to HIV-infected pregnant women at two different dosages:

* Group 1 (standard dosage): 200/50 mg lopinavir/r, 2 tablets every 12 hours, plus two nucleoside analogs.
* Group 2 (increased dosage): 200/50 mg lopinavir/r, 2 tablets every 12 hours until the end of the second trimester of gestation (24 weeks) and 3 tablets every 12 hours in the third trimester (from 25 weeks on), plus two nucleoside analogs.

Treatment will be initiated at any time between 14 and 30 weeks of gestation and will be maintained for at least 6 weeks after delivery.

The objectives are:

* To compare the pharmacokinetic parameters of the standard and increased dosage of the tablet formulation of lopinavir/r during pregnancy.
* To determine whether the standard and/or increased dosage of the tablet formulation of lopinavir/r during pregnancy confers the same exposure to the drug as that observed in the same women after the end of pregnancy and in historic controls.
* To evaluate the transplacental passage of lopinavir/r based on the ratio between the serum concentration in maternal blood at the time of delivery and in cord blood of the two drug dosages (standard and increased) administered during pregnancy.
* To evaluate the tolerability of the two lopinavir/r dosages (standard and increased) during pregnancy.
* To describe the vertical transmission rate of HIV to the children of the pregnant women included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent and wish to participate in the study, documented by signing the specific informed consent form (ICF) of the study.
* Age of 18 years or older.
* Pregnancy documented by urine or blood examination or ultrasound.
* Gestational age of 14 to 30 weeks calculated by ultrasound, obstetric examination or date of last menstruation, depending on what is considered to be more exact by the medical investigator.
* HIV infection documented by two serological tests using different methods or analysis of HIV viral load with a positive result.
* No use of antiretroviral drugs at the time of diagnosis of pregnancy (previous prophylaxis and treatment are allowed).
* Intention to continue the treatment of the study for at least 6 weeks after delivery.

Exclusion Criteria:

* History of hypersensitivity to lopinavir or ritonavir.
* Need for the concomitant use of contraindicated drugs in combination with lopinavir/ritonavir.
* Any condition that, in the opinion of the medical researchers, impairs the participation in and fulfillment of the procedures of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of the tablet formulation of lopinavir/r | Second and third pregnancy trimester and 6 weeks after delivery

SECONDARY OUTCOMES:
Ratio between the serum concentration of lopinavir/r in maternal blood and in cord blood | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Marilia S Oliveira, MD, Principal Investigator — IPEC - Oswaldo Cruz Foundation; Beatriz J Grinsztejn, MD, Principal Investigator — IPEC - Oswaldo Cruz Foundation; Eduardo W Barroso, MD, Principal Investigator — IPEC - Oswaldo Cruz Foundation; Valdilea G Veloso-Santos, MD, Principal Investigator — IPEC - Oswaldo Cruz Foundation; José Henrique S Pilotto, MD, Principal Investigator — Hospital Geral de Nova Iguaçu (HGNI)
Locations (3):
- Brazil (3):
  - Hospital Geral de Nova Iguaçu (HGNI), Nova Iguaçu, Rio de Janeiro
  - Hospital dos Servidores do Estado, Rio de Janeiro, Rio de Janeiro
  - Instituto de Pesquisa Clínica Evandro Chagas, Rio de Janeiro, Rio de Janeiro

REFERENCES:
- [Derived] Santini-Oliveira M, Estrela Rde C, Veloso VG, Cattani VB, Yanavich C, Velasque L, Torres TS, Marins LM, Pilotto JH, Joao EC, Goncalves JC, Grinsztejn B. Randomized clinical trial comparing the pharmacokinetics of standard- and increased-dosage lopinavir-ritonavir coformulation tablets in HIV-positive pregnant women. Antimicrob Agents Chemother. 2014 May;58(5):2884-93. doi: 10.1128/AAC.02599-13. Epub 2014 Mar 10. PMID 24614377